CLINICAL TRIAL: NCT00380042
Title: Feasibility Study of the Safety and Effectiveness of Cortical Stimulation for Subjects With Major Depressive Disorder
Brief Title: Assessment of the Safety and Effectiveness of Cortical Stimulation in Subjects With Major Depressive Disorder
Acronym: PROSPECT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated as a result of the dissolution of the Sponsor.
Sponsor: Northstar Neuroscience (Industry)
Responsible Party: VP Clinical Affairs, Northstar Neuroscience
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: V0479
Record Dates: First submitted 2006-09-21; First posted 2006-09-25 (Estimated); Last update posted 2009-12-31 (Estimated); Status verified 2008-09

CONDITIONS: Depression; Depressive Disorder
Keywords: Cortical Electrical Stimulation; Treatment Resistant Depression; Major Depressive Disorder
MeSH Terms: conditions — Depression; Depressive Disorder; Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Stimulation (Active Comparator)
  Interventions: Device: Cortical Stimulation
- Sham (Sham Comparator)
  Interventions: Device: Sham

INTERVENTIONS:
Device: Cortical Stimulation — Cortical stimulation of prefrontal cortex
  Other Names: Renova Cortical Stimulation System; Northstar Depression Treatment System (DTS)
  Arms: Active Stimulation
Device: Sham — Sham stimulation
  Arms: Sham

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of cortical stimulation to the cerebral cortex of subjects who have suffered from treatment-resistant depression and have failed routine attempts at controlling their depression.

DETAILED DESCRIPTION:
Major depressive disorders are the most common of all psychiatric disorders. The World Health Organization estimates that 340 million people worldwide suffer from an episode of major depression each year, accounting for 4.4% of the overall global disease burden. In the United States, about 9.5% or 19 million people are affected by a depressive disorder, with a lifetime risk of about 17% for a major depressive disorder.

While depression can be effectively treated in the majority of patients by medication and psychotherapy, up to 20% of patients fail to respond. Electroconvulsive Therapy (ECT) is effective in approximately 70% of cases where antidepressant medications do not provide sufficient relief of symptoms. However, as many as 20-50% of the people who respond well to a course of ECT relapse within 6 months, therefore, periodic maintenance therapy is often required.

For those patients who are resistant to the therapies noted above, more invasive approaches have been used, including Vagus Nerve Stimulation (VNS) and more recently Deep Brain Stimulation (DBS).

Direct cortical stimulation of the cortex via an implanted device system may provide long lasting benefit with minimal side effects. The current study seeks to assess in a feasibility study the safety and efficacy of stimulating the prefrontal cortex in patients with major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Current major depressive episode (MDE) lasting for at least two years, or at least 4 lifetime MDEs with the current episode lasting for at least one year
* Severe depression at study entry defined as a minimum score of 20 on the Hamilton Depression Rating Scale
* Failed response to at least four different antidepressant treatments

Exclusion Criteria:

* Axis I psychiatric diagnoses including schizophrenia, bipolar disorder, panic disorder, obsessive compulsive disorder, or evidence of global cognitive impairment
* An Axis II diagnoses of either: a) borderline personality disorder, or b) histrionic personality disorder
* Electroconvulsive therapy within 6 months prior to enrollment
* Known need of electroconvulsive therapy while the investigational device is implanted
* History of seizure disorder or status epilepticus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2006-09; Primary Completion 2007-10 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS28) | 8 weeks after implant surgery

SECONDARY OUTCOMES:
10-item Montgomery-Asberg Depression Rating Scale (MADRS) | 8 weeks after implant surgery

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: Click here for more information about this study: Cortical Stimulation for Depression — http://clinicaltrials.gov/ct2/show/NCT00380042